CLINICAL TRIAL: NCT06184828
Title: Pilot Study of Whole Blood Transfusion for Trauma Brain Injury (TBI)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Martin A Schreiber, MD, M.D., F.A.C.S., F.C.C.M., Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25989
Record Dates: First submitted 2023-12-07; First posted 2023-12-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exchange Transfusion, Whole Blood

STUDY DESIGN:
Intervention Model Description: Pilot, single center, and a randomized 1:1 trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Blood Transfusion (Experimental): Transfusion of whole blood units
  Interventions: Biological: Whole blood transfusion
- Blood Component Transfusion (Active Comparator): Transfusion of blood components units
  Interventions: Biological: Blood components transfusion

INTERVENTIONS:
Biological: Whole blood transfusion — The transfusion of whole blood units
  Arms: Whole Blood Transfusion
Biological: Blood components transfusion — The transfusion of blood components units rather than whole blood
  Arms: Blood Component Transfusion

SUMMARY:
Our goal is to perform a pilot, single center study to evaluate the efficacy of whole blood (WB) in subjects with TBI, intracranial hemorrhage, and anemia compared to blood component therapy.

DETAILED DESCRIPTION:
Both whole blood and blood components are given as standard-of-care based on the blood products available. If enrolled in this study, patients will be randomized 1:1 to receive either whole blood or blood components first. They will continue to receive blood products based on their assigned group. If they require more blood product than is available, they will cross over to the other group so they can continue to receive the transfusions needed for treatment.

The primary endpoint for this study would be improvement in coagulopathy pre and post intervention. Additionally, we will evaluate hemorrhagic progression of the intracranial bleed (HPIB), as measured by follow-up CT scan ordered over the first 24-hour post intervention (which is standard of care).

The secondary outcomes parameters would include intracranial pressure measurements (if performed), survival to discharge, safety and tolerability of Whole Blood administration in the TBI population, coagulation parameters and total blood product use, Glasgow Coma Scale (GCS) 24 hours post-injury, in-hospital mortality, and patient's discharge status (Glasgow Outcome Score Extended and disposition to home versus extended care facility).

Patients who decide to take part in the study, will have 26 mL of blood drawn (about 2 tablespoons) once before and once after blood transfusion for a total of 52 mL (about 4 tablespoons) of blood drawn, a CT scan at admission and at 24hour of blood transfusion, and information will be gathered from their medical record during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years and older
* Head CT with presence of intracranial bleeding
* Required transfusion of whole blood (WB) or red blood cells (RBC)

Exclusion Criteria:

* Patients with non-survivable injuries (expected to die within 24-hours of injury)
* Fixed and dilated pupils
* Patients requiring a massive transfusion protocol activation
* Receipt of 2 units of WB or RBCs prior to enrollment
* Known prisoners
* Known pregnancy

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality and Morbidity | Up to 30 days after hospital admission
  The primary outcome for this study would be Glasgow Outcome Coma Scale score at discharge.

SECONDARY OUTCOMES:
Improvement in Coagulopathy | Up to 30 days after hospital admission
  The secondary outcome for this study would be improvement in coagulopathy pre and post intervention. We will evaluate hemorrhagic progression of the intracranial bleed (HPIB), as measured by follow-up CT scan ordered over the first 24-hour post intervention (which is standard of care).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napolitano L. Cumulative risks of early red blood cell transfusion. J Trauma. 2006 Jun;60(6 Suppl):S26-34. doi: 10.1097/01.ta.0000199979.95789.17. No abstract available. PMID 16763477
- [Background] Timmons SD. The life-saving properties of blood: mitigating cerebral insult after traumatic brain injury. Neurocrit Care. 2006;5(1):1-3. doi: 10.1385/NCC:5:1:1. PMID 16960286
- [Background] Corwin HL, Carson JL. Blood transfusion--when is more really less? N Engl J Med. 2007 Apr 19;356(16):1667-9. doi: 10.1056/NEJMe078019. No abstract available. PMID 17442910
- [Background] Reiles E, Van der Linden P. Transfusion trigger in critically ill patients: has the puzzle been completed? Crit Care. 2007;11(3):142. doi: 10.1186/cc5936. PMID 17583592